CLINICAL TRIAL: NCT05317078
Title: Phase 1 First-In-Human Study to Explore the Safety, Tolerability, and Pharmacokinetics of AMG 794 in Participants With Claudin 6-positive Advanced/Metastatic Non-small Cell Lung Cancer, Epithelial Ovarian Cancer, and Other Malignant Solid Tumor Indications
Brief Title: A Phase 1 Safety, Tolerability, and Pharmacokinetics Study of AMG 794 With Claudin 6-positive Non-small Cell Lung Cancer, Epithelial Ovarian Cancer, and Other Malignant Solid Tumor Indications
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategic decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20210007
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Non-squamous Non-small Cell Lung Cancer; Epithelial Ovarian Cancer; Claudin 6-positive Advanced/Metastatic Malignant Solid Tumors
Keywords: Malignant solid tumors; Claudin 6-positive; AMG 794; CLDN6
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: AMG 794 (Experimental): Participants were planned to receive the lowest dose (Dose A), as a short-term IV infusion on Cycle 1 Day 1, with an increased dose on Cycle 1 Day 3 (Dose C) and Cycle 1 Day 8 (Dose E). After reaching the highest planned dose for the cohort (Dose E), participants continued to receive short-term IV infusions on Cycle 1 Day 15, then QW thereafter in 28-day cycles. Due to early study termination, participants only received Dose A on Cycle 1 Day 1 and Dose C on Cycle 1 Day 3.
  Interventions: Drug: AMG 794
- Cohort 1a: AMG 794 (Experimental): Participants were planned to receive the lowest dose (Dose A), as a short-term IV infusion on Cycle 1 Day 1, with an increased dose on Cycle 1 Day 8 (Dose B) and Cycle 1 Day 15 (Dose D). After reaching the highest planned dose for the cohort (Dose D), participants continued to receive short-term IV infusions QW thereafter in 28-day cycles.
  Interventions: Drug: AMG 794

INTERVENTIONS:
Drug: AMG 794 — Short-term intravenous (IV) infusion.

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of AMG 794 in adult participants and to determine the optimal biological active dose (OBD), at or below the maximum tolerated dose (MTD) with MTD 1 as the maximum tolerated starting dose and MTD 2 as the maximum tolerated target dose.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening:

* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 -1.
* Participants with histologically or cytologically documented malignant solid tumor diseases expressing claudin-6 (CLDN6) including but not limited to NSCLC, EOC, testicular germ cell cancer, uterine endometrial cancer, or triple negative breast cancer, and the cancer is at least either locally advanced or metastatic at pre-screening.
* Participant has provided informed consent prior to initiation of any study specific activities/procedures.

Main study:

* Age ≥ 18 years.
* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* ECOG performance status of 0 to 1.
* Participants with histologically or cytologically documented malignant solid tumor diseases expressing CLDN6 including but not limited to NSCLC, EOC, testicular germ cell cancer, uterine endometrial cancer, or triple negative breast cancer, that is metastatic or unresectable at screening time point. Participants should have exhausted available SOC systemic therapy or should not be candidates for such available therapy.
* For participants enrolling in cohort 3 or higher dose cohort, available positive test result for CLDN6 expression resulting from testing of an available archival tissue sample in pre-screening or obtained from biopsy in a screening procedure. For participants enrolling in cohorts 1, 1a, or 2 during dose escalation, consent to provide archival or fresh tumor tissue slides for immunohistochemistry (IHC) assessment is sufficient and the enrolment is not dependent on availability of the CLDN6 expression test result.
* For dose expansion cohorts: Participants with at least 1 measurable lesion ≥ 10mm which has not undergone biopsy within 3 months of screening scan. This lesion cannot be biopsied at any time during the study.
* Life expectancy > 3 months.
* Adequate organ functions.

Exclusion Criteria:

Main study:

* Positive test for human immunodeficiency virus, hepatitis B or hepatitis C.
* History of other malignancy within the past 2 years.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection with 1 week prior to administration of a first dose of study treatment
* Evidence of new or growing central nervous system metastases, leptomeningeal disease, or spinal cord compression. Participants with known brain metastases may be eligible if they completed radiotherapy, surgery or stereotactic surgery for the brain metastases and do not present with neurological symptoms and/or have stable disease assessed by imaging within 4 weeks of signing consent to this study and not requiring acute corticosteroid therapy or steroid taper.
* Currently receiving treatment in another investigational device or drug study, or less than 4 weeks since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Anticancer therapies including radiotherapy, chemotherapy or molecularly targeted treatments or tyrosine kinase inhibitors within 2 weeks or 5 half-lives (whichever is longer) of administration of a first dose of study treatment; immunotherapies/monoclonal antibodies within 3 weeks of administration of a first dose of study treatment.
* Has had a major surgery within 4 weeks of administration of a first dose of study treatment (excluded: biopsies and central venous catheter insertion).
* Autoimmune disorders requiring chronic systemic steroid therapy or any other form of immunosuppressive therapy while on study, (e.g., ulcerative colitis, Crohn's disease). Recent or current use of inhaled steroids or physiological substitution in case of adrenal insufficiency is not exclusionary.
* Female participants who are of childbearing potential unwilling to use protocol-specified method of contraception, who are breastfeeding and/or planning to become pregnant.
* Male participants who have a female partner of childbearing potential who are unwilling to practice sexual abstinence or use protocol-specified contraception and/or who are unwilling to abstain from donating sperm.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Day 1 to Day 28
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to a maximum of 2 years
  Adverse events (AEs) are defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occur after study treatment administration will be recorded as TEAEs.
Number of Participants Who Experience a Treatment-related AE | Day 1 to a maximum of 2 years

SECONDARY OUTCOMES:
Minimum Efficacious Dose (MED) | Day 1 to a maximum of 2 years
  Defined as the first unconfirmed partial response (PR) or better.
Maximum Observed Serum Concentration (Cmax) of AMG 794 | Cycle 1 Day 1 to Cycle 6 Day 1 (28 day cycle length)
Minimum Observed Serum Concentration (Cmin) of AMG 794 | Cycle 1 Day 1 to Cycle 6 Day 1 (28 day cycle length)
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval of AMG 794 | Cycle 1 Day 1 to Cycle 6 Day 1 (28 day cycle length)
Confirmed objective response (OR) | Day 1 to a maximum of 2 years
  Defined as best overall response [BOR] of complete response [CR] or PR based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Confirmed OR | Day 1 to a maximum of 2 years
  Defined as immune BOR (iBOR) of immune CR (iCR) or immune PR (iPR) based on Immune RECIST (iRECIST).
Cancer Antigen (CA) 125 Response | Day 1 to a maximum of 2 years
  CA 125 response will be analyzed in the Ovarian Cancer Analysis Set, defined as all participants with a primary tumor type of ovarian cancer who are enrolled and receive at least 1 dose of AMG 794.
Duration of Response | Day 1 to a maximum of 2 years
  Defined as the time from the first documentation of OR until the first documentation of disease progression or death due to any cause, whichever occurs first.
Time to Progression | Day 1 to a maximum of 2 years
  Defined as the time from enrollment until the first documentation of radiological disease progression.
Progression-free Survival (PFS) | Day 1 to a maximum of 2 years
  Defined as the time from enrollment until the first documentation of radiologic disease progression or death due to any cause, whichever occurs first.
1-year Overall Survival (OS) | 1 year
2-year OS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Cabrini Hospital, Malvern, Victoria
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com